CLINICAL TRIAL: NCT00452790
Title: A Phase 3, Randomised, Active-Controlled, Double-Blind Trial Evaluating the Safety, Tolerability and Immunogenicity of a 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants Given With Routine Paediatric Vaccinations in India
Brief Title: Study Evaluating 13-valent Pneumococcal Conjugate Vaccine in Healthy Infants in India
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Wyeth (Registry Contact: Clinical Trial Registry Specialist), Wyeth
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 6096A1-011
Record Dates: First submitted 2007-03-23; First posted 2007-03-27 (Estimated); Results first posted 2010-11-15 (Estimated); Last update posted 2011-03-24 (Estimated); Status verified 2011-03

CONDITIONS: Pneumococcal Infections
Keywords: Vaccines, Pneumococcal
MeSH Terms: conditions — Pneumococcal Infections | interventions — Heptavalent Pneumococcal Conjugate Vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- A (Experimental)
  Interventions: Biological: 13-valent Pneumococcal Conjugate Vaccine
- B (Active Comparator)
  Interventions: Biological: 7 valent pneumococcal conjugate vaccine

INTERVENTIONS:
Biological: 13-valent Pneumococcal Conjugate Vaccine — 1 dose at 6, 10, 14 weeks and 12 months of age
  Arms: A
Biological: 7 valent pneumococcal conjugate vaccine — 1 dose at 6, 10, 14 weeks and 12 months of age
  Arms: B

SUMMARY:
The purpose of this study is to assess the safety, tolerability and immunogenicity of a 13-valent pneumococcal conjugate vaccine (13vPnC) compared to Prevenar (7vPnC), when given concomitantly with routine paediatric vaccinations in India.

ELIGIBILITY:
Inclusion Criteria

1. Healthy infants aged 6 weeks (42-72 days) at time of enrolment
2. Available for the entire study period

Exclusion Criteria

1. Previous vaccination with pneumococcal, diphtheria, tetanus, pertussis or Hib vaccines
2. A previous anaphylactic reaction to any vaccine or vaccine-related component
3. Contraindication to vaccination with pneumococcal, Hib, diphtheria, tetanus, pertussis, polio, hepatitis B or measles vaccines

Ages: 42 Days to 72 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 708 (Actual)
Dates: Start 2007-06; Primary Completion 2009-10 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (9):
- India (9):
  - Sector-12, Chandigarh
  - Sector-32 B, Chandigarh
  - Bangalore, Karnataka
  - Mumbai, Maharashtra
  - Pune, Maharashtra
  - Rajinder Nagar, New Delhi
  - Ludhiana, Punjab
  - Chennai, Tamil Nadu
  - Vellore, Tamil Nadu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 708 participants were enrolled and 709 were randomized into the study. One infant in the 13vPnC group was randomly assigned twice because of technical difficulties with the first random assignment. Though this infant participated in the study only once, both random assignments were included in the 354 participants in the 13vPnC group.
Groups:
- 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC), administered intramuscularly, at 6, 10 and 14 weeks of age (infant series) and 12 months of age (toddler dose). During the infant series, 13vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, whole cell pertussis; H influenzae type b and hepatitis B vaccine (DTP-Hib-HBV); and a commercially available oral polio vaccine (OPV).
- 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 6, 10 and 14 weeks of age (infant series) and 12 months of age (toddler dose). During the infant series, 7vPnC was co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, whole cell pertussis; H influenzae type b and hepatitis B vaccine (DTP-Hib-HBV); and a commercially available oral polio vaccine (OPV).
Period: Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 354 | 355
Vaccinated Dose 1 | 353 | 353
Vaccinated Dose 2 | 300 | 300
Vaccinated Dose 3 | 221 | 218
Completed | 219 | 214
Not Completed | 135 | 141
Not completed — Clinical hold - consent withdrawn | 118 | 123
Not completed — Parent/legal guardian request | 8 | 6
Not completed — Failed to return | 4 | 1
Not completed — Protocol Violation | 1 | 3
Not completed — Lost to Follow-up | 2 | 2
Not completed — Adverse Event | 1 | 2
Not completed — Other reasons | 1 | 2
Not completed — Investigator request | 0 | 1
Not completed — Death | 0 | 1
Period: After Infant Series
Arm/Group | 13vPnC | 7vPnC
Started | 219 | 214
Completed | 198 | 200
Not Completed | 21 | 14
Not completed — Investigator request | 10 | 10
Not completed — Adverse Event | 4 | 1
Not completed — Parent/legal guardian request | 1 | 3
Not completed — Lost to Follow-up | 4 | 0
Not completed — Failed to return | 1 | 0
Not completed — Other reasons | 1 | 0
Period: Toddler Dose
Arm/Group | 13vPnC | 7vPnC
Started | 198 | 200
Completed | 198 | 198
Not Completed | 0 | 2
Not completed — Failed to return | 0 | 1
Not completed — Parent/legal guardian request | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 13vPnC | 7vPnC | Total
Number analyzed (Participants) | 354 | 355 | 709
Age Continuous [Mean (Standard Deviation); unit: months] | 1.6 (0.3) | 1.6 (0.2) | 1.6 (0.3)
Age Continuous [Mean (Standard Deviation); unit: weeks] | 7.1 (1.1) | 7.2 (1.1) | 7.1 (1.1)
Sex/Gender, Customized [Number; unit: participants]
  Male | 184 | 186 | 370
  Female | 169 | 169 | 338
  Unknown | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving a Predefined Antibody Level of Greater Than or Equal to 0.35 Micrograms (Mcg)/mL, 1 Month After the Infant Series.
Description: Percentage of participants achieving a predefined antibody level of greater than or equal to 0.35 mcg/mL along with the corresponding O'Brien-Fleming-adjusted, exact, 2-sided 95% confidence interval (CI) for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F and 19 A) are presented.
Time Frame: 1 month after the infant series (18 weeks of age)
Population: Evaluable immunogenicity population: had treatments as randomized at all 3 doses, blood drawn within specified timeframes, had at least 1 valid and determinate assay result for the proposed analysis, and no major protocol violations. n=number of participants with determinate IgG antibody concentration for the specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 206 | 196
Percentage of participants
  Common serotypes - serotype 4 (n= 203, 192) | 97.0 [93.6 to 98.9] | 97.9 [94.7 to 99.4]
  Common serotypes - serotype 6B (n= 196,194) | 84.7 [78.8 to 89.5] | 87.1 [81.5 to 91.5]
  Common serotypes - serotype 9V (n= 204,195) | 92.6 [88.1 to 95.8] | 94.4 [90.1 to 97.2]
  Common serotypes - serotype 14 (n= 185,186) | 91.4 [86.3 to 95.0] | 93.5 [89.0 to 96.6]
  Common serotypes - serotype 18C (n= 204,188) | 95.1 [91.1 to 97.6] | 93.1 [88.4 to 96.3]
  Common serotypes - serotype 19F (n= 200,188) | 95.0 [91.0 to 97.6] | 94.7 [90.4 to 97.4]
  Common serotypes - serotype 23F (n= 202,186) | 90.1 [85.1 to 93.9] | 89.2 [83.8 to 93.3]
  Additional serotypes - serotype 1 (n= 206,195) | 96.6 [93.1 to 98.6] | 0.5 [0.0 to 2.8]
  Additional serotypes - serotype 3 (n= 201,187) | 87.6 [82.1 to 91.8] | 2.1 [0.6 to 5.4]
  Additional serotypes - serotype 5 (n= 201,185) | 85.1 [79.3 to 89.7] | 24.3 [18.3 to 31.2]
  Additional serotypes - serotype 6A (n= 200,191) | 90.0 [84.9 to 93.8] | 36.1 [29.3 to 43.4]
  Additional serotypes - serotype 7F (n= 203,192) | 98.0 [95.0 to 99.5] | 2.6 [0.8 to 6.0]
  Additional serotypes - serotype 19 A (n= 204,190) | 99.5 [97.3 to 100.0] | 84.7 [78.8 to 89.6]

2. Other Pre Specified Outcome: Geometric Mean Concentration (GMC) for Serotype-specific Pneumococcal Immunoglobulin G (IgG) Antibody, 1 Month After the 3-Dose Infant Series
Description: Antibody GMC as measured in mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding O'Brien-Fleming-adjusted, 2-sided 95% CIs were calculated.
Time Frame: 1 month after the 3-dose infant series (18 weeks of age)
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 206 | 196
mcg/mL
  Common serotypes - serotype 4 (n= 203,192) | 2.19 [1.95 to 2.46] | 2.58 [2.26 to 2.95]
  Common serotypes - serotype 6B (n= 196,194) | 1.45 [1.20 to 1.75] | 1.56 [1.28 to 1.89]
  Common serotypes - serotype 9V (n= 204,195) | 1.34 [1.19 to 1.50] | 1.46 [1.28 to 1.65]
  Common serotypes - serotype 14 (n= 185,186) | 2.84 [2.35 to 3.43] | 2.39 [1.98 to 2.90]
  Common serotypes - serotype 18C (n= 204,188) | 1.61 [1.42 to 1.82] | 1.70 [1.47 to 1.96]
  Common serotypes - serotype 19F (n= 200,188) | 2.25 [1.97 to 2.56] | 2.47 [2.11 to 2.89]
  Common serotypes - serotype 23F (n= 202,186) | 1.38 [1.18 to 1.60] | 1.46 [1.25 to 1.70]
  Additional serotypes - serotype 1 (n= 206,195) | 1.95 [1.72 to 2.22] | 0.03 [0.03 to 0.04]
  Additional serotypes - serotype 3 (n= 201,195) | 0.80 [0.72 to 0.90] | 0.05 [0.05 to 0.06]
  Additional serotypes - serotype 5 (n= 201,195) | 0.93 [0.82 to 1.06] | 0.20 [0.18 to 0.23]
  Additional serotypes - serotype 6A (n= 200,195) | 1.44 [1.25 to 1.66] | 0.28 [0.25 to 0.31]
  Additional serotypes - serotype 7F (n= 203,195) | 2.27 [2.05 to 2.33] | 0.06 [0.05 to 0.06]
  Additional serotypes - serotype 19A (n= 204,195) | 2.76 [2.46 to 3.10] | 0.74 [0.66 to 0.82]

3. Primary Outcome: Percentage of Participants Achieving a Predefined Antibody Level for Concomitant Vaccine Pertussis Antigens (Pertussis Toxoid [PT], Filamentous Hemagglutinin [FHA], Pertactin [PRN]), 1 Month After the Infant Series.
Description: Percentage of participants achieving a predefined antibody level (measured in enzyme-linked immunosorbent assay [ELISA] units per mL [EU/mL]) along with the corresponding O'Brien-Fleming-adjusted, exact, 2-sided 95% CI for concomitant antigens pertussis (PT, FHA and PRN) are presented.
Time Frame: 1 month after the infant series (18 weeks of age)
Population: Evaluable immunogenicity population: had treatments as randomized at all 3 doses, blood drawn within specified timeframes, had at least 1 valid and determinate assay result for the proposed analysis, and no major protocol violations.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 206 | 196
Percentage of participants
  PT >=0.975 EU/mL | 100.0 [98.2 to 100.0] | 100.0 [98.1 to 100.0]
  FHA >=3.91 EU/mL | 100.0 [98.2 to 100.0] | 100.0 [98.1 to 100.0]
  PRN >=6 EU/mL | 92.7 [88.2 to 95.9] | 95.9 [92.1 to 98.2]

4. Secondary Outcome: Percentage of Participants Achieving a Predefined Antibody Level of Greater Than or Equal to 0.35 Mcg/mL, 1 Month After the Toddler Dose.
Description: Percentage of participants achieving a predefined antibody level of greater than or equal to 0.35 mcg/mL along with the corresponding exact, 2-sided 95% CI for the 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 5, 6A, 7F and 19 A) are presented.
Time Frame: 1 month after the toddler dose (13 months of age)
Population: Evaluable immunogenicity population: had treatments as randomized at all 4 doses, blood drawn within specified timeframes, had at least 1 valid and determinate assay result for the proposed analysis, and no major protocol violations. n=number of participants with determinate IgG antibody concentration for the specified serotype.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 193 | 196
Percentage of participants
  Common serotypes - serotype 4 (n= 193, 196) | 100.0 [98.1 to 100.0] | 100.0 [98.1 to 100.0]
  Common serotypes - serotype 6B (n= 192,195) | 100.0 [98.1 to 100.0] | 99.5 [97.2 to 100.0]
  Common serotypes - serotype 9V (n= 193,196) | 99.5 [97.1 to 100.0] | 99.5 [97.2 to 100.0]
  Common serotypes - serotype 14 (n= 193,196) | 99.5 [97.1 to 100.0] | 99.5 [97.2 to 100.0]
  Common serotypes - serotype 18C (n= 193,196) | 99.5 [97.1 to 100.0] | 99.0 [96.4 to 99.9]
  Common serotypes - serotype 19F (n= 193,196) | 97.9 [94.8 to 99.4] | 98.0 [94.9 to 99.4]
  Common serotypes - serotype 23F (n= 193,196) | 98.4 [95.5 to 99.7] | 99.5 [97.2 to 100.0]
  Additional serotypes - serotype 1 (n= 193,196) | 98.4 [95.5 to 99.7] | 3.1 [1.1 to 6.6]
  Additional serotypes - serotype 3 (n= 193,196) | 90.2 [85.1 to 94.0] | 12.9 [8.5 to 18.4]
  Additional serotypes - serotype 5 (n= 192,196) | 100.0 [98.1 to 100.0] | 74.3 [67.4 to 80.5]
  Additional serotypes - serotype 6A (n= 193,196) | 100.0 [98.1 to 100.0] | 92.8 [88.2 to 96.0]
  Additional serotypes - serotype 7F (n= 193,196) | 99.0 [96.3 to 99.9] | 9.8 [6.0 to 14.9]
  Additional serotypes - serotype 19 A (n= 193,196) | 100.0 [98.1 to 100.0] | 98.5 [95.5 to 99.7]

5. Other Pre Specified Outcome: GMC for Serotype-specific Pneumococcal IgG Antibody, 1 Month After the Toddler Dose
Description: Antibody GMC as measured in mcg/mL for 7 common pneumococcal serotypes (serotypes 4, 6B, 9V, 14, 18C, 19F, and 23F) and 6 additional pneumococcal serotypes specific to 13vPnC (Serotypes 1, 3, 5, 6A, 7F, and 19A) are presented. GMC (13vPnC) and corresponding 2-sided 95% CIs were presented.
Time Frame: 1 month after toddler dose (13 months of age)
Population: as for outcome 4
Measure: Geometric Mean (95% Confidence Interval); unit: mcg/mL
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 193 | 196
mcg/mL
  Common serotypes - serotype 4 (n= 193, 196) | 5.33 [4.69 to 6.04] | 5.85 [5.13 to 6.68]
  Common serotypes - serotype 6B (n= 192, 195) | 12.24 [10.60 to 14.13] | 11.60 [9.95 to 13.53]
  Common serotypes - serotype 9V (n= 193,196) | 3.01 [2.68 to 3.37] | 3.33 [2.96 to 3.75]
  Common serotypes - serotype 14 (n= 193,196) | 10.59 [9.21 to 12.18] | 10.95 [9.41 to 12.74]
  Common serotypes - serotype 18C (n= 193,196) | 2.63 [2.33 to 2.97] | 2.98 [2.65 to 3.34]
  Common serotypes - serotype 19F (n= 193,196) | 8.38 [7.11 to 9.87] | 5.65 [4.84 to 6.58]
  Common serotypes - serotype 23F (n= 193,196) | 4.27 [3.66 to 4.98] | 5.31 [4.66 to 6.04]
  Additional serotypes - serotype 1 (n= 193,196) | 5.10 [4.39 to 5.92] | 0.04 [0.04 to 0.05]
  Additional serotypes - serotype 3 (n= 193,196) | 0.91 [0.81 to 1.03] | 0.09 [0.08 to 0.11]
  Additional serotypes - serotype 5 (n= 192,196) | 3.58 [3.20 to 4.00] | 0.64 [0.55 to 0.75]
  Additional serotypes - serotype 6A (n= 193,196) | 8.13 [7.11 to 9.28] | 1.87 [1.62 to 2.17]
  Additional serotypes - serotype 7F (n= 193,196) | 4.81 [4.27 to 5.42] | 0.06 [0.05 to 0.08]
  Additional serotypes - serotype 19A (n= 193,196) | 14.12 [12.45 to 16.01] | 3.56 [3.14 to 4.05]

6. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Infant Series Dose 1 (6 Weeks of Age)
Description: Local reactions were reported using an electronic diary. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and erythema were scaled as Any (induration or erythema present); Mild (0.5 cm to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after the dose 1 of the infant series (6 weeks of age)
Population: Safety population: all participants who received dose 1 of the infant series vaccination (6 weeks of age). n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 353 | 353
Percentage of participants
  Tenderness: Any (n= 347,347) | 62.5 | 59.7
  Tenderness: Significant (n= 341,343) | 42.2 | 40.5
  Induration: Any (n= 339,342) | 21.5 | 22.5
  Induration: Mild (n= 338,340) | 19.2 | 19.1
  Induration: Moderate (n= 331,338) | 4.8 | 5.6
  Induration: Severe (n= 329,336) | 0.0 | 0.0
  Erythema: Any (n= 333,339) | 12.6 | 13.3
  Erythema: Mild (n= 333,338) | 11.4 | 11.8
  Erythema: Moderate (n= 330,337) | 1.5 | 1.8
  Erythema: Severe (n= 329,336) | 0.0 | 0.0
  Any of the above (n= 349,348) | 66.8 | 65.2
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-any within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.483, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-significant within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.698, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-any within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.782, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-mild within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-moderate within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.729, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Induration-Severe within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Erythema-Any within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.819, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-mild within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.904, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Erythema-Moderate within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-severe within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any local reaction (tenderness, induration and erythema) within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.690, Fisher Exact

7. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Infant Series Dose 2 (10 Weeks of Age)
Description: as for outcome 6
Time Frame: Within 4 days after the dose 2 of the infant series (10 weeks of age)
Population: Safety population: all participants who received the first 2 doses of the infant series vaccination (10 weeks of age).n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 300 | 300
Percentage of participants
  Tenderness: Any (n= 284,282) | 44.4 | 44.0
  Tenderness: Significant (n= 278,279) | 26.6 | 28.0
  Induration: Any (n= 281,278) | 20.6 | 18.7
  Induration: Mild (n= 281,277) | 16.7 | 16.2
  Induration: Moderate (n= 273,272) | 5.1 | 4.0
  Induration: Severe (n= 273,271) | 0.0 | 0.0
  Erythema: Any (n= 275,280) | 13.8 | 17.9
  Erythema: Mild (n= 275,279) | 13.1 | 15.8
  Erythema: Moderate (n= 273,273) | 1.5 | 2.9
  Erythema: Severe (n= 273,271) | 0.0 | 0.0
  Any of the above (n= 285,286) | 51.6 | 53.1
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-any within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.933, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-significant within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.776, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-any within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.596, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-mild within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.909, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-moderate within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.683, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-severe within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-any within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.203, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Erythema-Mild within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.399, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-moderate within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.382, Fisher Exact
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-severe within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any Local reaction (tenderness, induration, erythema) within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.738, Fisher Exact

8. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Infant Series Dose 3 (14 Weeks of Age)
Description: Local reactions were reported using an electronic diary by the parent/legal guardian. Tenderness was scaled as Any (tenderness present); Significant (present and interfered with limb movement). Induration and erythema were scaled as Any (induration and erythema present); Mild (0.5 cm to 2.0 cm); Moderate (2.5 to 7.0 cm); Severe (> 7.0 cm). Participants may be represented in more than 1 category.
Time Frame: Within 4 days after the dose 3 of the infant series (14 weeks of age)
Population: Safety population: all participants who received all 3 doses of the infant series vaccination (14 weeks of age).n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 221 | 218
Percentage of participants
  Tenderness: Any (n= 204,200) | 37.3 | 38.0
  Tenderness: Significant (n= 199,196) | 24.1 | 23.5
  Induration: Any (n= 198,195) | 17.2 | 13.8
  Induration: Mild (n= 196,195) | 15.8 | 11.8
  Induration: Moderate (n= 193,193) | 2.6 | 3.6
  Induration: Severe (n= 191,193) | 0.0 | 0.0
  Erythema: Any (n= 192,195) | 10.4 | 9.7
  Erythema: Mild (n= 192,195) | 10.4 | 9.2
  Erythema: Moderate (n= 191,193) | 0.0 | 0.5
  Erythema: Severe (n= 191,193) | 0.0 | 0.0
  Any of the above (n= 206,202) | 43.2 | 42.1
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-any within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.918, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-significant within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.906, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-any within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.404, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-mild within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.305, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-moderate within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.771, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-severe within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-any within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.867, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-mild within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.735, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-moderate within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-severe within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any Local Reaction (tenderness, induration, erythema) within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.842, Fisher Exact

9. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Local Reactions: Toddler Dose (12 Months of Age)
Description: as for outcome 8
Time Frame: Within 4 days after the toddler dose (12 months of age)
Population: Safety population: all participants who received toddler dose vaccination(after 12 months). n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 198 | 200
Percentage of participants
  Tenderness: Any (n= 174,176) | 29.9 | 30.7
  Tenderness: Significant (n= 171,170) | 15.8 | 17.1
  Induration: Any (n= 173,176) | 19.7 | 17.6
  Induration: Mild (n= 170,175) | 15.9 | 14.9
  Induration: Moderate (n= 170,171) | 5.3 | 7.6
  Induration: Severe (n= 167,169) | 0.0 | 0.0
  Erythema: Any (n= 174,176) | 14.9 | 14.2
  Erythema: Mild (n= 172,175) | 12.2 | 10.9
  Erythema: Moderate (n= 169,170) | 3.6 | 4.1
  Erythema: Severe (n= 167,169) | 0.0 | 0.0
  Any of the above (n= 177,178) | 36.7 | 41.0
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-any within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.908, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of tenderness-significant within 4 days of the toddler dose, dose 4(12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.772, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-any within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.681, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-mild within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.881, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-moderate within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.509, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of induration-severe within 4 days of the toddler dose (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-any within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.880, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-mild within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.739, Fisher Exact
Statistical Analysis 9: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-moderate within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 10: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of erythema-severe within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 11: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any local reaction (tenderness, induration, erythema) within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.446, Fisher Exact

10. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Infant Series Dose 1 (6 Weeks of Age)
Description: Systemic events (any fever >=38 degrees Celsius [C], decreased appetite, irritability, increased sleep, decreased sleep) were reported using an electronic diary. Participants may be represented in more than 1 category.
Time Frame: Within 4 days after the dose 1 of the infant series (6 weeks of age)
Population: Safety population: all participants who received at least dose 1 of the infant series vaccination (after 6 weeks. n=number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 353 | 353
Percentage of participants
  Fever >=38 but <=39 degrees C (n= 313,324) | 19.8 | 21.6
  Fever >39 but <=40 degrees C (n= 309,322) | 2.3 | 1.2
  Fever >40 degrees C (n= 309,322) | 0.3 | 0.9
  Decreased appetite (n= 343,347) | 55.7 | 55.9
  Irritability (n= 345,347) | 83.2 | 79.8
  Increased sleep (n= 338,342) | 40.8 | 36.8
  Decreased sleep (n= 336,343) | 55.7 | 56.0
  Any systemic event (n= 350,348) | 94.3 | 90.8
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >=38 but <=39 degrees C within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.625, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >39 but <=40 degrees C within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.375, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >40 degrees C within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.624, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of decreased appetite within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of irritability within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.282, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Increased sleep within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.307, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of decreased sleep within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.939, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any systemic event (fever, decrease in appetite, irritability, increased or decreased sleep) within 4 days of the infant series dose 1 (6 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.085, Fisher Exact

11. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Infant Series Dose 2 (10 Weeks of Age)
Description: as for outcome 10
Time Frame: Within 4 days after the dose 2 of the infant series (10 weeks of age)
Population: Safety population: all participants who received dose 2 of the infant series vaccination (10 weeks of age); n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 300 | 300
Percentage of participants
  Fever >=38 but <=39 degrees C (n= 263,249) | 10.3 | 15.3
  Fever >39 but <=40 degrees C (n= 259,247) | 0.8 | 0.4
  Fever >40 degrees C (n= 259,247) | 0.0 | 0.4
  Decreased appetite (n= 281,282) | 48.0 | 46.5
  Irritability (n= 290,291) | 70.7 | 69.8
  Increased sleep (n= 285,275) | 33.7 | 26.9
  Decreased sleep (n= 282,286) | 37.9 | 46.9
  Any systemic event (n= 294,297) | 80.6 | 80.5
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >= 38 but <= 39 degrees C within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.111, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >39 but <= 40 degrees C within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >40 degrees C within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.488, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Decreased appetite within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.736, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Irritability within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.856, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Increased sleep within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.098, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Decreased sleep within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.034, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of Any systemic event (fever, decrease in appetite, irritability, increased or decreased sleep) within 4 days of the infant series dose 2 (10 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact

12. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Infant Series Dose 3 (14 Weeks of Age)
Description: as for outcome 10
Time Frame: Within 4 days after the dose 3 of the infant series (14 weeks of age)
Population: Safety population: all participants who received dose 3 of the infant series vaccination (14 weeks of age).n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 221 | 218
Percentage of participants
  Fever >=38 but <=39 degrees C (n= 181,172) | 7.7 | 14.0
  Fever >39 but <=40 degrees C (n= 179,170) | 0.0 | 0.0
  Fever >40 degrees C (n= 179,171) | 0.0 | 0.6
  Decreased appetite (n= 202,200) | 42.1 | 41.0
  Irritability (n= 208,208) | 64.4 | 67.3
  Increased sleep (n= 199,195) | 20.1 | 20.5
  Decreased sleep (n= 205,201) | 42.4 | 36.8
  Any systemic event (n= 213,209) | 75.1 | 78.5
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >= 38 but <= 39 degrees C within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.085, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >39 but <= 40 degrees C within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >40 degrees C within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.489, Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of decreased appetite within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.840, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of irritability within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.605, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of increased sleep within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of decreased sleep within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.265, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any systemic event (fever, decrease in appetite, irritability, increased or decreased sleep) within 4 days of the infant series dose 3 (14 weeks of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.422, Fisher Exact

13. Other Pre Specified Outcome: Percentage of Participants With Pre-specified Systemic Events: Toddler Dose (12 Months of Age)
Description: as for outcome 10
Time Frame: Within 4 days after the toddler dose(12 months of age)
Population: Safety population: all participants who received toddler dose vaccination (12 months of age).n= number of participants reporting yes for at least 1 day or no for all days for each treatment group respectively.
Measure: Number; unit: Percentage of participants
Arm/Group | 13vPnC | 7vPnC
Number analyzed (Participants) | 198 | 200
Percentage of participants
  Fever >=38 but <=39 degrees C (n= 161,154) | 5.6 | 6.5
  Fever >39 but <=40 degrees (n= 160,152) | 0.6 | 0.0
  Fever >40 degrees C (n= 160,152) | 0.0 | 0.0
  Decreased appetite (n= 174,179) | 28.7 | 24.6
  Irritability (n= 174,183) | 38.5 | 35.0
  Increased sleep (n= 171,170) | 12.3 | 9.4
  Decreased sleep (n= 172,178) | 22.7 | 27.0
  Any systemic event (n= 179,186) | 54.7 | 52.7
Statistical Analysis 1: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >= 38 but <= 39 degrees within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.815, Fisher Exact
Statistical Analysis 2: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >39 but <= 40 degrees within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p > 0.99, Fisher Exact
Statistical Analysis 3: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of fever >40 degrees C within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; Fisher Exact
Statistical Analysis 4: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of decreased appetite within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.401, Fisher Exact
Statistical Analysis 5: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of irritability within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.511, Fisher Exact
Statistical Analysis 6: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of increased sleep within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.487, Fisher Exact
Statistical Analysis 7: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of decreased sleep within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.388, Fisher Exact
Statistical Analysis 8: Comparison: 13vPnC vs 7vPnC; Difference in incidence rates of any systemic event fever, decrease in appetite, irritability, increased or decreased sleep) within 4 days of the toddler dose, dose 4 (12 months of age) reported in the 13vPnC group relative to the incidence rates in the 7vPnC group. No hypothesis testing was performed. The analysis is descriptive; Test type: Superiority or Other; p = 0.753, Fisher Exact

ADVERSE EVENTS:
Time Frame: Baseline through 1 month after last study vaccination (13 Months). Local reactions and systemic events assessed within 4 days of dose: Infant Series Dose 1=6 weeks of age; Dose 2=10 weeks of age; Dose 3=14 weeks of age; Toddler Dose=12 months of age.
Description: Safety population = all randomized subjects with at least 1 dose of study treatment. An Adverse Event (AE) term may be reported as both a serious and non-serious AE, but are distinct events. AE may = serious for 1 subject and = non-serious for another subject or subject may have experienced both a serious and non-serious episode of the same event
Groups:
- Infant Series 13vPnC: Participants received 1 single 0.5 mL dose of 13-valent pneumococcal conjugate vaccine (13vPnC), administered intramuscularly, at 6, 10 and 14 weeks of age (infant series), co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, whole cell pertussis; H influenzae type b and hepatitis B vaccine (DTP-Hib-HBV); and a commercially available oral polio vaccine (OPV).
- Infant Series 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 6, 10 and 14 weeks of age (infant series), co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, whole cell pertussis; H influenzae type b and hepatitis B vaccine (DTP-Hib-HBV); and a commercially available oral polio vaccine (OPV).
- After the Infant Series 13vPnC: Participants received 1 single 0.5 mL dose of 13vPnC, administered intramuscularly, at 6, 10 and 14 weeks of age (infant series), co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, whole cell pertussis; H influenzae type b and hepatitis B vaccine (DTP-Hib-HBV); and a commercially available oral polio vaccine (OPV). AEs were collected from approximately 1 month after Dose 3 to the Toddler dose.
- After the Infant Series 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 6, 10 and 14 weeks of age (infant series), co-administered with a commercially available combination vaccine containing: diphtheria, tetanus, whole cell pertussis; H influenzae type b and hepatitis B vaccine (DTP-Hib-HBV); and a commercially available oral polio vaccine (OPV). AEs were collected from approximately 1 month after Dose 3 to the Toddler dose.
- Toddler Dose 13vPnC: Participants received 1 single 0.5 mL dose of 13vPnC, administered intramuscularly, at 12 months of age (toddler dose).
- Toddler Dose 7vPnC: Participants received 1 single 0.5 mL dose of 7vPnC, administered intramuscularly, at 12 months of age (toddler dose).
Arm/Group | Infant Series 13vPnC | Infant Series 7vPnC | After the Infant Series 13vPnC | After the Infant Series 7vPnC | Toddler Dose 13vPnC | Toddler Dose 7vPnC
Serious Adverse Events (participants affected / at risk) | 8/353 | 6/353 | 8/353 | 11/353 | 4/198 | 1/200
Other Adverse Events (participants affected / at risk) | 330/353 | 316/353 | 5/353 | 9/353 | 98/198 | 98/200
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Infant Series 13vPnC (N=353) | Infant Series 7vPnC (N=353) | After the Infant Series 13vPnC (N=353) | After the Infant Series 7vPnC (N=353) | Toddler Dose 13vPnC (N=198) | Toddler Dose 7vPnC (N=200)
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 1 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Bronchiolitis (Infections and infestations) | 2 | 4 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 3 | 0 | 1 | 1 | 1 | 0
Meningitis bacterial (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0
Heart disease congenital (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Hepatosplenomegaly (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 4 | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Lower respiratory tract infection viral (Infections and infestations) | 0 | 0 | 2 | 1 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 2 | 0 | 0 | 0
Dysentery (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Viral myocarditis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 2 | 1 | 0 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Breath holding (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Infant Series 13vPnC (N=353) | Infant Series 7vPnC (N=353) | After the Infant Series 13vPnC (N=353) | After the Infant Series 7vPnC (N=353) | Toddler Dose 13vPnC (N=198) | Toddler Dose 7vPnC (N=200)
Ventricular extrasystoles (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0 | 0 | 0 | 0
Otorrhoea (Ear and labyrinth disorders) | 1 | 0 | 0 | 0 | 0 | 0
Eye discharge (Eye disorders) | 2 | 1 | 0 | 0 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 21 | 26 | 1 | 0 | 1 | 3
Vomiting (Gastrointestinal disorders) | 4 | 6 | 0 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Infantile colic (Gastrointestinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Flatulence (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Perianal erythema (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Injection site pain (General disorders) | 75 | 70 | 0 | 0 | 0 | 0
Injection site swelling (General disorders) | 55 | 57 | 0 | 0 | 0 | 0
Pyrexia (General disorders) | 29 | 21 | 0 | 0 | 2 | 6
Injection site erythema (General disorders) | 12 | 12 | 0 | 0 | 0 | 0
Injection site nodule (General disorders) | 5 | 12 | 0 | 0 | 0 | 0
Irritability (General disorders) | 1 | 3 | 0 | 0 | 0 | 0
Tenderness (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinitis (Infections and infestations) | 47 | 37 | 0 | 3 | 1 | 4
Upper respiratory tract infection (Infections and infestations) | 39 | 45 | 2 | 2 | 11 | 6
Nasopharyngitis (Infections and infestations) | 11 | 17 | 0 | 1 | 1 | 2
Gastroenteritis (Infections and infestations) | 8 | 5 | 0 | 0 | 2 | 3
Lower respiratory tract infection (Infections and infestations) | 5 | 2 | 1 | 1 | 0 | 0
Bronchiolitis (Infections and infestations) | 4 | 2 | 0 | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 2 | 3 | 0 | 0 | 0 | 0
Bronchopneumonia (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0
Viral infection (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 1
Acarodermatitis (Infections and infestations) | 0 | 2 | 0 | 0 | 1 | 0
Omphalitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Viral diarrhoea (Infections and infestations) | 2 | 0 | 0 | 0 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 1
Abscess neck (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Body tinea (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Fungal infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Impetigo (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Oral candidiasis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Otitis candidiasis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract infection viral (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Viral rash (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Limb injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Crying (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Umbilical granuloma (Pregnancy, puerperium and perinatal conditions) | 0 | 1 | 0 | 0 | 0 | 0
Penile adhesion (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 37 | 40 | 0 | 2 | 5 | 6
Upper airway obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 1 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 2 | 2 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 2 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 0 | 0 | 0
Acne infantile (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Macrocephaly (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 1 | 0 | 0
Tuberculosis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Rickets (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0
Febrile convulsion (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 2
Phimosis (Congenital, familial and genetic disorders) | 0 | 0 | 0 | 0 | 1 | 0
Allergy to arthropod bite (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetitie (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 1
Tenderness (any) (Skin and subcutaneous tissue disorders) | 217/347 | 207/347 | 0/0 | 0/0 | 52/174 | 54/176 — Infant Series Dose 1 and Toddler Dose; Tenderness (any) = present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 126/284 | 124/282 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; tenderness (any) = present at site of vaccination.
Tenderness (any) (Skin and subcutaneous tissue disorders) | 76/204 | 76/200 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; tenderness (any)= present at site of vaccination.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 144/341 | 139/343 | 0/0 | 0/0 | 27/171 | 29/170 — Infant Series Dose 1 and Toddler Dose; Tenderness (significant) = present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 74/278 | 78/279 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Tenderness (significant) = present and interfered with limb movement.
Tenderness (significant) (Skin and subcutaneous tissue disorders) | 48/199 | 46/196 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Tenderness (significant) = present and interfered with limb movement.
Induration (any) (Skin and subcutaneous tissue disorders) | 73/339 | 77/342 | 0/0 | 0/0 | 34/173 | 31/176 — Infant Series Dose 1 and Toddler Dose; Induration (any) = present at site of vaccination.
Induration (any) (Skin and subcutaneous tissue disorders) | 58/281 | 52/278 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (any) = present at site of vaccination.
Induration (any) (Skin and subcutaneous tissue disorders) | 34/198 | 27/195 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (any) = present at site of vaccination.
Induration (mild) (Skin and subcutaneous tissue disorders) | 65/338 | 65/340 | 0/0 | 0/0 | 27/170 | 26/175 — Infant Series Dose 1 and Toddler Dose; Induration (mild) = 0.5 to 2.0 centimeters (cm)
Induration (mild) (Skin and subcutaneous tissue disorders) | 47/281 | 45/277 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (mild) = 0.5 to 2.0 cm
Induration (mild) (Skin and subcutaneous tissue disorders) | 31/196 | 23/195 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (mild) = 0.5 to 2.0 cm
Induration (moderate) (Skin and subcutaneous tissue disorders) | 16/331 | 19/338 | 0/0 | 0/0 | 9/170 | 13/171 — Infant Series Dose 1 and Toddler Dose; Induration (moderate) = 2.5 to 7.0 cm
Induration (moderate) (Skin and subcutaneous tissue disorders) | 14/273 | 11/272 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (moderate) = 2.5 to 7.0 cm
Induration (moderate) (Skin and subcutaneous tissue disorders) | 5/193 | 7/193 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (moderate) = 2.5 to 7.0 cm
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/329 | 0/336 | 0/0 | 0/0 | 0/167 | 0/169 — Infant Series Dose 1 and Toddler Dose; Induration (severe) >7.0 cm
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/273 | 0/271 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Induration (severe) >7.0 cm
Induration (severe) (Skin and subcutaneous tissue disorders) | 0/191 | 0/193 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Induration (severe) >7.0 cm
Erythema (any) (Skin and subcutaneous tissue disorders) | 42/333 | 45/339 | 0/0 | 0/0 | 26/174 | 25/176 — Infant Series Dose 1 and Toddler Dose; Erythema (any) = present at site of vaccination.
Erythema (any) (Skin and subcutaneous tissue disorders) | 38/275 | 50/280 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (any) = present at site of vaccination
Erythema (any) (Skin and subcutaneous tissue disorders) | 20/192 | 19/195 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (any) = present at site of vaccination
Erythema (mild) (Skin and subcutaneous tissue disorders) | 38/333 | 40/338 | 0/0 | 0/0 | 21/172 | 19/175 — Infant Series Dose 1 and Toddler Dose; Erythema (mild) = 0.5 to 2.0 cm
Erythema (mild) (Skin and subcutaneous tissue disorders) | 36/275 | 44/279 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (mild) = 0.5 to 2.0 cm
Erythema (mild) (Skin and subcutaneous tissue disorders) | 20/192 | 18/195 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (mild) = 0.5 to 2.0 cm
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 5/330 | 6/337 | 0/0 | 0/0 | 6/169 | 7/170 — Infant Series Dose 1 and Toddler Dose; Erythema (moderate) = 2.5 to 7.0 cm
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 4/273 | 8/273 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (moderate) = 2.5 to 7.0 cm
Erythema (moderate) (Skin and subcutaneous tissue disorders) | 0/191 | 1/193 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (moderate) = 2.5 to 7.0 cm
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/329 | 0/336 | 0/0 | 0/0 | 0/167 | 0/169 — Infant Series Dose 1 and Toddler Dose; Erythema (severe) >7.0 cm
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/273 | 0/271 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Erythema (severe) >7.0 cm
Erythema (severe) (Skin and subcutaneous tissue disorders) | 0/191 | 0/193 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Erythema (severe) >7.0 cm
Fever ≥ 38 degrees Celsius [C] but ≤ 39 degrees C (General disorders) | 62/313 | 70/324 | 0/0 | 0/0 | 9/161 | 10/154 — Infant Series Dose 1 and Toddler Dose; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 27/263 | 38/249 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever ≥ 38 degrees C but ≤ 39 degrees C (General disorders) | 14/181 | 24/172 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever ≥ 38 degrees C but ≤ 39 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 7/309 | 4/322 | 0/0 | 0/0 | 1/160 | 0/152 — Infant Series Dose 1 and Toddler Dose; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 2/259 | 1/247 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 39 degrees C but ≤ 40 degrees C (General disorders) | 0/179 | 0/170 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 39 degrees C but ≤ 40 degrees C
Fever > 40 degrees C (General disorders) | 1/309 | 3/322 | 0/0 | 0/0 | 0/160 | 0/152 — Infant Series Dose 1 and Toddler Dose; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/259 | 1/247 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Fever > 40 degrees C
Fever > 40 degrees C (General disorders) | 0/179 | 1/171 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Fever > 40 degrees C
Decreased appetite (General disorders) | 191/343 | 194/347 | 0/0 | 0/0 | 50/174 | 44/179 — Infant Series Dose 1 and Toddler Dose; Decreased appetite
Decreased appetite (General disorders) | 135/281 | 131/282 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased appetite
Decreased appetite (General disorders) | 85/202 | 82/200 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased appetite
Irritability (General disorders) | 287/345 | 277/347 | 0/0 | 0/0 | 67/174 | 64/183 — Infant Series Dose 1 and Toddler Dose; Irritability
Irritability (General disorders) | 205/290 | 203/291 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Irritability
Irritability (General disorders) | 134/208 | 140/208 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Irritability
Increased sleep (General disorders) | 138/338 | 126/342 | 0/0 | 0/0 | 21/171 | 16/170 — Infant Series Dose 1 and Toddler Dose; Increased sleep
Increased sleep (General disorders) | 96/285 | 74/275 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Increased sleep
Increased sleep (General disorders) | 40/199 | 40/195 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Increased sleep
Decreased sleep (General disorders) | 187/336 | 192/343 | 0/0 | 0/0 | 39/172 | 48/178 — Infant Series Dose 1 and Toddler Dose; Decreased sleep
Decreased sleep (General disorders) | 107/282 | 134/286 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 2; Decreased sleep
Decreased sleep (General disorders) | 87/205 | 74/201 | 0/0 | 0/0 | 0/0 | 0/0 — Infant Series Dose 3; Decreased sleep

LIMITATIONS AND CAVEATS:
Geometric Mean Concentration Outcome Measures were identified as secondary analysis in the study protocol, but are included to maintain consistency with other postings for this program.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.